CLINICAL TRIAL: NCT03732625
Title: Neuropsyquiatric Evolution After Introduction of Raltegravir QD in Substitution of Dolutegravir: NEAR QD Study
Acronym: NEARQD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FIMHCSBR-2017
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-12

CONDITIONS: HIV Infections
Keywords: HIV infection; neuropsychological adverse effects; Raltegravir
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Mutation, Missense

STUDY DESIGN:
Intervention Model Description: Multicenter, open, non-randomized pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Raltegravir (Experimental): Raltegravir (RAL) x 2 600mg QD (Total 1200mg QD)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — DTG will be replaced by Raltegravir (RAL) 1200 QD, maintaining the other two drugs that constituted the triple therapy established before the inclusion of the patient in the study.
  Other Names: Substitution

SUMMARY:
Open, multicenter, non randomized, single arm, pilot trial.

DETAILED DESCRIPTION:
Open, multicenter, non randomized, single arm, pilot trial. The study is aimed at patients infected with HIV in triple antiretroviral therapy based on Dolutegravir (DTG) who experience neuropsychological adverse effects related to the treatment. After signing the informed consent, DTG will be replaced by Raltegravir (RAL) 1200 QD, maintaining the other two drugs that constituted the triple therapy established before the inclusion of the patient in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Infection with chronic HIV-1.
* On triple therapy antiretroviral therapy based on abacavir/lamivudine (ABC/3TC) or tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) or tenofovir alafenamide/emtricitabine (TAF/FTC), whose third component is DTG in a dose of 50 mg / day.
* Presence of neuropsychiatric symptoms (insomnia, sleep disturbances, reduced concentration, dizziness, headaches, depression, restlessness or nervousness) with an intensity ≥ 2 on the DAIDS scale.
* Written informed consent to participate in the study.

Exclusion criteria:

* Pregnant women, nursing or of childbearing age who want to get pregnant.
* Concomitant use of any medication with potential risk of interaction with the therapy under study.
* Intolerance, hypersensitivity or previous resistance to the therapy under study or presence of any contraindication of it.
* Subjects in therapy with immunosuppressants or chemotherapy with cytotoxics, including interferon and interleukin-2 at the time of their inclusion in the study.
* Abuse of alcohol or any other substance that may interfere with adherence to treatment.
* Subjects who are participating in any other clinical study with the exception of those in which the treatment under study has been suspended for more than 12 weeks.
* AIDS event at the time of diagnosis of HIV infection or in the 3 months prior to its inclusion
* Any other clinical condition or previous treatment that makes the subject unsuitable for the study or that compromises their ability to comply with the treatment dosing requirements.
* History of mental illness or diagnosis of neuropsychological symptoms prior to the use of DTG.
* Presence of genotypic mutations that confer resistance to ABC, TDF / TAF, 3TC or FTC.
* Chronic liver disease in the cirrhosis phase (either by ultrasound criteria or fibroscan ≥ 14.5 KPa)
* Consumption of tobacco ≥ 20 cigarettes / day.

Additional Exclusion Criteria (for patients recruited at the Costa del Sol Hospital in Marbella only):

* History or diagnosis of claustrophobia, or inability to lie flat on the back inside the positron emission tomograph or MRI chamber for a period of 20 minutes.
* Contraindication to perform an MRI, including the presence of a cardiac pacemaker or other electronic device or ferromagnetic metallic foreign bodies in vulnerable positions evaluated by a standard questionnaire prior to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate improvement in neuropsychiatric symptoms at 12 weeks (Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events) | 12 weeks
  Evaluate improvement in neuropsychiatric symptoms: grade 1 to 4 of DAIDS scale. higher values represent a worse outcome

SECONDARY OUTCOMES:
Neuropsychiatric symptoms | 24 weeks
  Presence and Intensity of neuropsychiatric symptoms (visual scale 0 to 10)
Interruptions of the medication for any reason | 24 weeks
  Interruptions of the medication due to adverse effects, virological failure, or any other reason
Change in quality of life (WHOQoL-bref questionnaire) | 24 weeks
  World Health Organization Quality of Life: 1-100 in 4 domains. 100 best score
Variation of the result in the Hospital, Anxiety and Depression (HAD) scale | 24 weeks
  Hospital, anxiety and depression: 0 y 7 indicates no case, between 8 & 10 indicates doubtful case and scores of 11 and above are possibly anxiety and depression cases.
Variation of the result on the Pittsburgh Sleep Quality Index (PSQI) scale | 24 weeks
  Pittsburgh Sleep Quality Index: Score 0 to 21 points. "0" indicates ease of sleeping and "21" severe difficulty in all areas.
Variation of the result in the Epworth scale | 24 weeks
  Diurnal drowsiness: If score is less than 6 points, daytime sleepiness is low or absent; between 7 and 8, is in the average of the population and if it is higher than 9 its drowsiness is excessive.
Variation of the result in the COLUMBIA-SUICIDE SEVERITY RATING (CSSR) scale | 24 weeks
  COLUMBIA-SUICIDE SEVERITY RATING SCALE: progressive score depending of each question answer
Magnetic Resonance Imagigng (MRI) analysis for 10 of the patients recruited at the Costa del Sol Hospital (pilot subestudy) | 24 weeks
  * Identify patterns of different metabolic marker 18F-fluorodeoxyglucose (18F-FDG) uptake in patients suffering from central nervous system toxicity in relation to the use of Dolutegravir after replacement with Raltegravir.
  * Observe if the anatomic-functional pattern of these patients changes after the substitution of Dolutegravir by Raltegravir.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Olalla, PhD, Study Director — SAS
Locations (3):
- Spain (3):
  - Costa del Sol University Hospital, Marbella, Málaga
  - Clínic University Hospital, Barcelona
  - San Carlos Clinical Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No